CLINICAL TRIAL: NCT01573338
Title: Phase Ib / II Study of BAY 1000394 in Combination With Cisplatin / Etoposide or Carboplatin / Etoposide as First-line Therapy in Subjects With Extensive Disease Small Cell Lung Cancer
Brief Title: Clinical Study to Evaluate the Maximum Tolerated Dose of BAY1000394 When Given Together With Chemotherapy and the Effectiveness of This Combination Treatment in Shrinking a Specific Type of Lung Tumors (Small Cell Lung Cancer)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14858; 2011-004155-39 (EudraCT Number)
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Cyclin dependent kinases; Drug therapy, combination; Small cell lung carcinoma; Etoposide; Cisplatin; Carboplatin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — roniciclib; Etoposide; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): BAY1000394 will be administered in combination with chemotherapy (etoposide and cisplatin or carboplatin) for up to 6 cycles. BAY1000394 will continue beyond Cycle 6 of chemotherapy. Type of chemotherapy for each patient will be decided by the investigator case by case.
  Interventions: Drug: Roniciclib (BAY1000394); Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Roniciclib (BAY1000394) — oral administration twice daily in a 3 days on/ 4 days off schedule. Starting dose will be 2.5 mg bid and dose will be escalated or de-escalated depending on dose limiting toxicity.
Drug: Etoposide — 100 mg/m2 will be administered IV on Days 1, 2, and 3 of each 21 day cycle.
Drug: Cisplatin — 75 mg/m2 will be administered IV on Day 1 of each 21 day cycle after the etoposide infusion is complete.
Drug: Carboplatin — Carboplatin will be administered IV on Day 1 of each 21 day cycle. The dose of carboplatin will be determined for each cycle using the Calvert's formula, to yield an AUC of 5 (mg/mL) • min.

SUMMARY:
This is the first study where BAY1000394 is given in combination with chemotherapy: cisplatin / etoposide or carboplatin / etoposide. Patients with small cell lung cancer will be treated. Every patient will receive drug treatment, there is no placebo group. Different groups of patients will receive different dosages of BAY1000394 to determine the safety and maximum tolerated dose (MTD) of BAY1000394 in combination with chemotherapy. The dose of chemotherapy is the standard dose usually administered and will not change.

The study will also assess how the drug is metabolized by the body and changes in tumor size.

BAY1000394 will be given per mouth, twice a day for three days every week. Treatment will stop if the tumor continues to grow, if side effects occur which the patient can not tolerate or if the patients decides to exit treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged >/=18 years
* Histologically or cytologically confirmed, extensive disease SCLC
* At least 1 solid tumor lesion measurable by computer tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST 1.1. Subjects with non-measurable disease according to RECIST 1.1 can be included in the Phase Ib part of the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Life expectancy of at least 12 weeks
* Serum sodium >/=130 mmol/L

Exclusion Criteria:

* Prior systemic anticancer therapy
* Prior radiotherapy (local palliative radiotherapy is permitted)
* History of cardiac disease: congestive heart failure > NYHA Class II, unstable angina (anginal symptoms at rest), any episodes of angina or history of myocardial infarction, cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted), previous venous or arterial thrombotic events, pulmonary embolism
* Moderate or severe hepatic impairment, ie Child-Pugh class B or C
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-06-23 (Actual)

PRIMARY OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events collection | up to 3 years
tumor response - number of subjects with best tumor response that is achieved during or within 30 days after end of therapy | up to 3 years
Maximum Tolerated Dose (MTD) - measured by adverse event profile at the end of Cycle 1. MTD will be the highest dose level achieved during dose escalation where non or 1 of 6 subjects experience a dose limiting toxicity as defined in the protocol | up to 3 years
Maximum drug concentration in plasma after single dose administration(Cmax) of BAY1000394 | Cycle 1, Day 8 and Cycle 2, Day 1
Area under the concentration versus time curve from zero to infinity after single (first) dose(AUC) of BAY1000394 | Cycle 1, Day 8 and Cycle 2, Day 1

SECONDARY OUTCOMES:
Disease control rate (DCR) | From start of treatment of the first subject until 3 years later, assessed every 6 weeks
  number of patients with complete response, partial response or stable disease according to RECIST
Overall survival (OS) | From start of treatment of the first subject until 3 years later
  time (days) from date of first treatment to death due to any cause.
Time to progression (TTP) | From start of treatment of the first subject until 3 years later, assessed every 6 weeks
  time (days) from date of first treatment to first observed radiological disease progression
Progression-free survival (PFS) | From start of treatment of the first subject until 3 years later, assessed every 6 weeks
  time (days) from date of first treatment to first observed radiological disease progression or death
Duration of response (DOR) | From start of treatment of the first subject until 3 years later, assessed every 6 weeks
  time (days) from date of first radiological response to the date that progressive disease is first radiologically documented or death occurs
Stable disease (SD) | From start of treatment of the first subject until 3 years later, assessed every 6 weeks
  time (days) from date of first treatment to first observed radiological disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (3):
  - St Louis, Missouri
  - Buffalo, New York
  - Cleveland, Ohio
- France (3):
  - Caen
  - Marseille
  - Villejuif
- Seoul, South Korea

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/